CLINICAL TRIAL: NCT03001804
Title: Use of Lenalidomide (Revlimid®) in Combination With Dexamethasone in Untreated Non-transplantable Multiple Myeloma in Practice
Brief Title: Use Lenalidomide (Revlimid®) in Combination With Dexamethasone in Clinical Practice for the Treatment of Newly Diagnosed Multiple Myeloma (MM) Transplant Ineligible Patients
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-5013-MM-037
Record Dates: First submitted 2016-12-19; First posted 2016-12-23 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Revlimid; Lenalidomide; Non-transplantable
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: Lenalidomide 25mg or 10mg (reduced renal function 30 ≤ ClCr < 50mg/min) capsules by mouth (PO) on days 1 through 21 of a 28 day cycle and Dexamethasone 40mg PO (≤75 years) or 20mg (>75years) on Days 1, 8, 15, 22 of a 28 day cycle until progression or unacceptable toxicity
- Cohort B: Initial treatment (up to 8 cycles): Lenalidomide 25mg or 10mg (reduced renal function 30 ≤ ClCr < 50mg/min) capsule by mouth (PO) on day 1 through 14 of a 21 day cycle, Bortezomib 1.3mg/m2 s.c. on day 1, 4, 8, and 11 of a 21 day cycle, and Dexamethasone 20mg PO on days 1,2,4,5,8,9,11,12 of a 21 day cycle; Successive Treatment: Lenalidomide 25mg or 10mg (reduced renal function 30 ≤ ClCr < 50mg/min) capsules by mouth (PO) on days 1 through 21 of a 28 day cycle and Dexamethasone 40mg PO (≤75 years) or 20mg (>75years) on Days 1, 8, 15, 22 of a 28 day cycle until progression or unacceptable toxicity

SUMMARY:
The aim of this non-interventional study is to collect primarily the percentage of patients who receive the full dose of dexamethasone (20 or 40 mg orally once daily on days 1, 8, 15 and 22 of the repetitive 28-day cycles, 20 mg in >75 year old patients) in the registered indication under practice conditions.

DETAILED DESCRIPTION:
Multiple myeloma is still a persistent and life-threatening blood cancer that is characterised by tumour proliferation and suppression of the immune system. It is a rare but incurable disease. On average, multiple myeloma is diagnosed in people 65-74 years of age, and the majority of newly diagnosed patients may not be eligible for more aggressive treatment options such as high-dose chemotherapy with stem cell transplant. In February 2015 REVLIMID® (lenalidomide) was approved in combination with dexamethasone for the treatment of adult patients with previously untreated multiple myeloma who are not eligible for transplant. Furthermore, in May 2019 REVLIMID® was approved in combination with bortezomib and dexamethasone for the treatment of adult patients with previously untreated multiple myeloma who are not eligible for transplant.

Looking in more detail at the combination of lenalidomide and dexamethasone, the role and especially the most adequate and effective dosage of dexamethasone in long term use with lenalidomide is not clearly defined or well characterised It is therefore of great relevance to gain insights into the clinical practice and the routine of dexamethasone management and dosing in long term use with Revlimid.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Age ≥ 18 years
* Newly diagnosed Multiple Myeloma
* Not suitable for stem cell transplantation
* Appropriate methods of contraception according to the Risk Minimization Program (RMP)
* Adequate thrombosis prophylaxis

Exclusion Criteria:

* Pregnant and lactating females
* No other formal exclusion criteria according to most recent European Summary of Product Characteristics (SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for therapy of untreated multiple myeloma, where stem cell transplantation cannot be performed
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Number of patients receiving dexamethasone after 6 months of treatment | up to 2 years
  Number of patients receiving 20mg or 40mg dexamethasone on day 1, 8, 15, 22 of a 28 day cycle after 6 months of treatment

SECONDARY OUTCOMES:
Number of patients with Deep Venous Thrombosis (VTE) prophylaxis | up to 2 years
  Number of patients that receive VTE prophylaxis
Over all response rate (ORR) | up to 2 years
  Number of patients that achieve a response
Adverse Events (AEs) | up to 2 years
  Number of patients with an adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- Austria (12):
  - Landeskrankenhaus Kirchdorf, Kirchdorf
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Kepleruniversitätsklinikum GmbH, Hämatologie und Internistische Onkologie, Linz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Krankenhaus der Barmherzigen Schwestern Ried Innere Medizin 1, Ried
  - Landeskrankenhaus Steyr - Innere Medizin, Steyr
  - AKH, Innere Medizin I, Klinische Abteilung für Hämatologie und Hämostaseologie, Vienna
  - Klinische Abteilung für Hämatologie und Hämostaseologie, Vienna
  - St. Josef Krankenhaus, Vienna
  - Wilhelminenspital, 1. Med.Abteilung, Zentrum für Onkologie, Vienna
  - Salzkammergut-Klinikum Vöcklabruck Abteilung Innere Medizin, Vöcklabruck
  - LKH Wiener Neustadt, Innere Medizin, Wiener Neustadt